CLINICAL TRIAL: NCT05284799
Title: Phase 2a, Randomized, Double-blind (Double-dummy), Controlled, Parallel-group Study to Evaluate the Immunogenicity and the Safety of the Concomitant Administration of OVX836 Influenza Vaccine and a Quadrivalent Inactivated Influenza Vaccine Given Intramuscularly as 2 Separate Injections in the Same Arm, in Comparison to Co-administration of Quadrivalent Inactivated Influenza Vaccine and Placebo and to Co-administration of OVX836 and Placebo Given Intramuscularly in Healthy Subjects.
Brief Title: Immunogenicity and Safety of the Concomitant Administration of OVX836 and Quadrivalent Influenza Vaccine in Healthy Volunteers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: Northern Beaches Clinical Research (Unknown); Novotech (Australia) Pty Limited (Industry); Harmony Clinical Research BVBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-004
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2022-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Randomized assignment (1:1:1) into 3 groups of 60 subjects to receive:
  * First group: OVX836 480µg and Quadrivalent Inactivated Influenza Vaccine at commercial dose administered
  * Second group: Quadrivalent Inactivated Influenza Vaccine at commercial dose, concomitantly administered with placebo
  * Third group: OVX836 480µg, concomitantly administered with placebo
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OVX836 480µg + Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose (Experimental): OVX836: Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein of the incluenza virus. One single administration intramuscularly of 480µg dose on Day 1
  AND
  Fluarix® Tetra (GlaxoSmithKline Biologicals): Inactivated and purified split influenza vaccine.
  Interventions: Biological: OVX836 480µg; Biological: Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra)
- Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose + Placebo (Active Comparator): Fluarix® Tetra (GlaxoSmithKline Biologicals): Inactivated and purified split influenza vaccine.
  AND
  Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50mL. One single administration intrumuscularly of a 0.8mL dose on Day 1
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra); Biological: Placebo
- OVX836 480µg + Placebo (Placebo Comparator): OVX836: Adjuvant-free recombinant influenza candidate vaccine based on Nucleoprotein of the incluenza virus. One single administration intramuscularly of 480µg dose on Day 1
  AND
  Placebo Comparator: Saline solution (B. Braun Ecoflac Plus) Saline solution (NaCl 0,9%), B. Braun Ecoflac Plus 50mL. One single administration intrumuscularly of a 0.8mL dose on Day 1
  Interventions: Biological: OVX836 480µg; Biological: Placebo

INTERVENTIONS:
Biological: OVX836 480µg — One single administration intramuscularly at Day 1
  Arms: OVX836 480µg + Placebo; OVX836 480µg + Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose
Biological: Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) — One single administration intramuscularly at Day 1
  Arms: OVX836 480µg + Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose; Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose + Placebo
Biological: Placebo — One single administration intramuscularly at Day 1
  Arms: OVX836 480µg + Placebo; Quadrivalent Inactivated Influenza Vaccine (Fluarix® Tetra) at commercial dose + Placebo

SUMMARY:
The present study will evaluate the concomitant administration of a Quadrivalent Inactivated Influenza Vaccine with the highest dose level of OVX836 (480µg) tested in the clinic to date, for which the likelihood for interference with Quadrivalent Inactivated Influenza Vaccine is considered the highest.

DETAILED DESCRIPTION:
This trial is a Phase 2a, randomized, double-blind, controlled study in 180 adult subjects to compare the immunogenicity and the safety of the concomitant administration (given intramuscularly, in healthy subjects, as 2 separate injections in the same arm) of:

* OVX836 influenza vaccine and a Quadrivalent Inactivated Influenza Vaccine
* Quadrivalent Inactivated Influenza Vaccine and placebo
* OVX836 influenza vaccine and placebo

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Between the age of 18 and 55 years, inclusive.
4. Subjects who have fully been vaccinated with licensed Severe Acute Respiratory Syndrome Coronavirus-2 (COVID-19) vaccine(s) according to national recommendations for the corresponding population group, in vigor at the moment the study starts.
5. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.
6. Ability and technical possibility for completing an e-diary and ePRO.

Exclusion Criteria:

1. Subjects with a body mass index ≤19 kg/m² or ≥35 kg/m² on the day of vaccination.
2. Previous influenza vaccination within 6 months before the day of vaccination or planned to receive during the study duration.
3. Any known or suspected immunodeficient conditions.
4. Past or current history of significant autoimmune diseases, as judged by the Investigator.
5. Current history of uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases.
6. Known or suspected infection with human immunodeficiency virus, hepatitis C virus, or hepatitis B virus, based upon medical history or physical examination findings.
7. Female subjects: pregnant, breast-feeding or of childbearing potential without appropriate contraceptive methods in place for 2 months before enrolment, or with positive pregnancy test on the day of vaccination. Appropriate contraceptive methods are to be maintained until the end of the trial. Appropriate contraceptive methods are defined by the Clinical Trial Facilitation Group as follow: "Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable intrauterine device, intrauterine hormone-releasing system), bilateral tubal occlusion, vasectomized partner and/or sexual abstinence (refraining from heterosexual intercourse)."
8. Having received another vaccination within 3 months prior to the day of study vaccination with live attenuated vaccines, or within 1 month prior to the day of study vaccination with inactivated vaccines, except COVID-19 vaccine.
9. Planning to receive other vaccines during the first 28 days following the study vaccine administration, except COVID-19 vaccine.
10. Having received a COVID-19 vaccination within 2 weeks prior to the day of study vaccination.
11. Planning to receive COVID-19 vaccine during the first week (within 7 days) following the study vaccine administration. An interval of preferably 14 days is recommended. If for scheduling reasons, COVID-19 vaccine has to be given on Day 8, the vaccination should be administered after completion of the study procedures.
12. Administration of any investigational or non-registered drug or vaccine within 3 months prior to the administration of study vaccines, or planned administration of any such product during the whole study period.
13. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
14. Presence of an acute febrile illness on the day of vaccination (oral temperature >38.0°C, temporary exclusion criterion).
15. Past or current history of any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
16. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
17. Past (stopped less than 6 months before enrolment) or current history of alcohol or drug abuse, or current smoking habit above 10 cigarettes per day, or current vaping.
18. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 30 days before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, interferon, immunomodulators, allergy shots, as judged by the Investigator.
19. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to any component of either of the study vaccines, including to egg protein or to kanamycin.
20. Any contraindication to IM administration, as judged by the Investigator, including bleeding disorders such as hemophilia or anticoagulant therapy.
21. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
22. Subjects with tattoos in the deltoid region bilaterally, which might interfere with observation of local signs and symptoms or other adverse events at the injection sites. In case of tattoos on one side, injections of study vaccines should be performed in the contralateral arm.
23. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted, including children of newly composed families.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Number of seroconversion determined using Hemagglutination-Inhibition assay, for the four influenza strains contained in the Quadrivalent Influenza Vaccine. | At Day 29 versus pre-injection baseline (Day 1)
  Seroconversion is defined as a negative pre-vaccination Hemagglutination-Inhibition assay titer and post-vaccination Hemagglutination-Inhibition assay titer ≥1:40, or a fourfold increase in Hemagglutination-Inhibition assay titer between pre- and post-vaccination timepoints.
Proportion of subjects achieving a titer ≥1:40 at Day 29 determined using Hemagglutination-Inhibition assay, for the four influenza strains contained in the Quadrivalent Influenza Vaccine. | At Day 29
Number of Hemagglutination-Inhibition assay titers geometric mean ratios >2.5 for the four influenza strains contained in the Quadrivalent Influenza Vaccine. | At Day 29 versus pre-injection baseline (Day 1)
Proportion of subjects reporting solicited local (Injection site redness, Injection site swelling, Injection site pain) and systemic signs and symptoms (Fatigue, Headache, Arthralgia, Malaise, Myalgia, Fever) | During 7 days after vaccine administration
Proportion of subjects reporting unsolicited AEs | During 29 days after vaccine administration
Proportion of subjects with Influenza-Like-Illness cases | During the whole study duration, 180 days
Severity scores of Influenza-Like-Illness cases (as per Flu-PRO questionnaire) | During the whole study duration, 180 days
Proportion of subjects reporting Serious Adverse Events | During the whole study duration, 180 days

SECONDARY OUTCOMES:
Hemagglutination-Inhibition assay geometric mean titers for each of the four strains contained in the Quadrivalent Influenza Vaccine. | At Day 1 (pre-injection baseline) and Day 29
Cell-mediated immune response in terms of change of Nucleoprotein-specific T-cell frequencies in Peripheral Blood Mononuclear Cells, measured by Interferon Gamma Enzyme-Linked Immunospot Assay. | At Day 8 versus pre-injection baseline (Day 1)
Geometric Mean Titer of anti-Nucleoprotein immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum). | At Day 1, Day 8 and Day 29
Proportion of subjects with an increase (four-fold) in anti-Nucleoprotein Immunoglobulin G (Enzyme-Linked Immunosorbent Assay, serum) titer. | At Day 29 with respect to pre-injection baseline (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Aldrich, MBBS, Principal Investigator — Northern Beaches Clinical Research
Locations (1):
- Northern Beaches Clinical Research, Brookvale, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groth N, Bruhwyler J, Tourneur J, Piat E, Moris P, Le Vert A, Nicolas F. Safety and Immunogenicity of OVX836, a Nucleoprotein-Based Universal Influenza Vaccine, Co-Administered with Fluarix(R) Tetra, a Seasonal Hemagglutinin-Based Vaccine. Vaccines (Basel). 2025 May 23;13(6):558. doi: 10.3390/vaccines13060558. PMID 40573889